CLINICAL TRIAL: NCT01936103
Title: Effects of Intensive Statin Therapy on Left Ventricular Function for Patients With the First Acute Anterior Myocardial Infarction After Directly to Percutaneous Coronary Intervention.
Brief Title: Effects of Intensive Statin Treatment on Left Ventricular Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, MD, vice president, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NH-20120404
Record Dates: First submitted 2013-04-23; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-08

CONDITIONS: Acute Anterior Myocardial Infarction
Keywords: Acute anterior myocardial infarction; Percutaneous coronary stent implantation; Intensive statin therapy; Left ventricular function
MeSH Terms: conditions — Anterior Wall Myocardial Infarction | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard group (Active Comparator): patients in this group received standard statin treatment： Atorvastatin statins 20mg / night .
  Interventions: Drug: standard group
- intensive group (Experimental): patients in this group received intensive statin treatment： Admission atorvastatin statins the 80mg, after surgery，atorvastatin 40mg / night，and until 30 days after the operation , and thereafter 20mg / night .
  Interventions: Drug: intensive group

INTERVENTIONS:
Drug: standard group — standard statin treatment:Atorvastatin statins 20mg / night .
  Other Names: Lipitor
  Arms: standard group
Drug: intensive group — intensive statin treatment： Admission atorvastatin statins the 80mg, after surgery，atorvastatin 40mg / night，and until 30 days after the operation
  Other Names: intensive Lipitor
  Arms: intensive group

SUMMARY:
First acute anterior myocardial infarction in patients with primary PCI preoperative and postoperative 30 days intensive dose atorvastatin statin therapy compared with conventional -dose therapy , patients can improve left ventricular function , reduce major adverse cardiovascular events .

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. the first time clinical diagnosis of acute anterior myocardial infarction , the time of onset ≤ 12 hours ,intends underwent emergency PCI
3. informed consent

Exclusion Criteria:

1. Taking , or the need for long-term use of statins is greater than the initial dose
2. treated with PCI again within a mouth
3. active liver disease or liver dysfunction
4. the diagnosis of myopathy
5. severe renal insufficiency ( serum creatinine > 178umol / L )
6. Statin drug allergy or had a serious adverse reaction
7. severe aortic stenosis or mitral stenosis , hypertrophic obstructive cardiomyopathy , pericardial disease
8. pregnancy
9. malignancy or any other end-stage diseases result in a life expectancy of < 6 months
10. be participating in other clinical studies
11. not suitable for inclusion of the other cases
12. not treated with PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-05 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
left ventricular function | 30 days
  ultrasonic observation of left ventricular end-diastolic diameter
left ventricular function | 30 days
  ultrasonic observation of left ventricular end-systolic volume
left ventricular function | 30 days
  ultrasonic observation of left ventricular fractional shortening RWSI
left ventricular function | 30 days
  ultrasonic observation of the left ventricular ejection fraction
left ventricular function | 30 days
  ultrasonic observation of E/A

SECONDARY OUTCOMES:
the left ventricular function | 6 months
the left ventricular function | 1 year
plasma brain natriuretic peptide | 30days
plasma brain natriuretic peptide | 6 months
plasma brain natriuretic peptide | 1 year

OTHER OUTCOMES:
enzymes | 1 year
  the level of CK peak
Major adverse cardiac and cerebral events at 1 year | 1 year
  1 year after death, cardiac death , myocardial infarction , heart failure , cardiac causes hospitalization , revascularization combined endpoint of cerebrovascular events .
Aspartate aminotransferase (AST) | 1 year
  Aspartate aminotransferase (AST) returned to normal in the perioperative period
enzymes | 1 year
  CK-MB peak
enzymes | 1 year
  troponin (TnT)
enzymes | 1 year
  CK-MB peak time
Aspartate aminotransferase (AST) | 1 year
  any elevation> 3 times the proportion
alanine aminotransferase (ALT) | 1 year
  alanine aminotransferase (ALT)returned to normal in the perioperative period
alanine aminotransferase (ALT) | 1 year
  any elevation> 3 times the proportion

CONTACTS AND LOCATIONS:
Overall Officials: Geng Wang, Dr, Study Director — Shenyang Northern Hospital
Locations (1):
- Shenyang Northen Hospital, Shenyang, Liaoning, China